CLINICAL TRIAL: NCT04217239
Title: A Comparison of Short-term and Long- Term Outcomes Between Ivor-Lewis and McKeown Minimally Invasive Esophagectomy
Brief Title: A Comparison Between Ivor-Lewis and McKeown Minimally Invasive Esophagectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIE ZYP2
Record Dates: First submitted 2020-01-01; First posted 2020-01-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Esophageal Cancer
Keywords: Thoracoscopic; laparoscopic; esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivor-Lewis group (Experimental): minimally invasive esophagectomy (MIE) with intrathoracic anastomosis
  Interventions: Procedure: MIE Ivor- Lewis
- McKeown group (Active Comparator): minimally invasive esophagectomy (MIE) with cervical anastomosis
  Interventions: Procedure: MIE McKeown

INTERVENTIONS:
Procedure: MIE Ivor- Lewis — minimally invasive esophagectomy (MIE) with intrathoracic anastomosis
  Arms: Ivor-Lewis group
Procedure: MIE McKeown — minimally invasive esophagectomy (MIE) with cervical anastomosis
  Arms: McKeown group

SUMMARY:
Surgery is still the main treatment for esophageal cancer, however, the complication and mortality rate of open esophagectomy is high. As a result, the thoracoscopic- laparoscopic minimally invasive esophagectomy (MIE) was developed. The MIE mainly comprised two surgical approaches:

MIE McKeown approach (cervical anastomosis) and MIE Ivor-Lewis approach (intrathoracicanastomosis). The MIE with intrathoracic anastomosis (Ivor-Lewis) is increasingly used for the treatment of mid and lower esophageal cancers. Our study is trying to compare the safety, feasibility, and short-term and long- term outcomes between MIE Ivor-Lewis approach and MIE McKeown approach for the treatment of lower thoracic esophageal cancer and esophageal- gastric junction.

ELIGIBILITY:
Inclusion Criteria:

(I) Patients with clinically staged T1-3N0-2M0 tumors; good cardiopulmonary function;

(II) Patients with lower thoracic esophageal tumors and esophageal- gastric junction tumor;

(III) Patients without a previous history of cancer;

(IV) Patients without a previous history of neck or chest surgery;

Exclusion Criteria:

(I) cardiopulmonary function not good enough for surgery;

(II) Patients with hybrid MIE

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Overall postoperative complications | within one month
  Overall postoperative complication rates

SECONDARY OUTCOMES:
Operating time | 1 day
  Operating time in minutes
Lymph nodes harvested | 1 day
  Lymph nodes harvested in number
Blood loss | 1 day
  Blood loss in milliliter
Anastomotic leak | within one month
  Anastomotic leak in rate
Pulmonary complication | 1 month
  Pulmonary complication in rate
Anastomotic stenosis | within three months
  Anastomotic stenosis in rate
recurrent laryngeal nerve injury | within three months
  recurrent laryngeal nerve injury in rate
Chylothorax | within one month
  Chylothorax in rate
Cardiac arrhythmia | within one month
  Cardiac arrhythmia in rate
Laboratory findings | within 3 days
  Three-day postoperative laboratory findings including ALB, PA, Glob, etc.
Hospital stay | within 60 days
  Hospital stay in days
mortality | within 30 and 90 days
  mortality in rate
progression-free survival | within 5 years
  progression-free survival in rate

CONTACTS AND LOCATIONS:
Locations (1):
- Yunpeng Zhao, Jinan, Shandong, China

REFERENCES:
- [Derived] Zhao Y, Shan L, Peng C, Cong B, Zhao X. Learning curve for minimally invasive oesophagectomy of oesophageal cancer and survival analysis. J Cardiothorac Surg. 2021 Nov 10;16(1):328. doi: 10.1186/s13019-021-01712-7. PMID 34758861